CLINICAL TRIAL: NCT05731557
Title: ACE, Resilience, and Substance Use Disorder: Maternal and Baby Outcomes in the First Year of Life
Status: Completed | Type: Observational
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Alla Kushnir, Associate Professor of Pediatrics, Principal Investigator, The Cooper Health System
Other Study IDs: 20-025
Record Dates: First submitted 2022-03-07; First posted 2023-02-16 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Adverse Childhood Experiences

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to understand maternal factors, including ACE and 7Cs Tool scores, and how they contribute to the health of mothers and their infant. The study will evaluate whether or not the outcomes of maternal and baby health can be identified early through the Adverse Childhood Experiences (ACE) questionnaire, 7Cs Tool questionnaire, and Maternal Health Questionnaire.

Additionally, the study will ask questions regarding current maternal social factors that could influence labor and delivery.

DETAILED DESCRIPTION:
Adverse Childhood Experiences (ACEs) are traumatic or life-threatening events that occurred to an individual during the ages 0-17 and are measured with the ACE Score questionnaire. These experiences include being a victim of physical and sexual abuse, neglect, and exposure to household dysfunction such as parental substance abuse or incarceration1. Multiple studies have shown that the number of ACEs an individual experiences correlates with his or her risk in developing chronic health issues such as diabetes, asthma, and hypertension later in life 2-4. In addition, ACEs correlate with a higher risk of engaging in risky behaviors such as substance use5. A recent survey conducted by the Substance Abuse and Mental Health Services Administration (SAMHSA) showed that 5.4% of pregnant mothers had used illicit drugs including marijuana, opioids, and cocaine in the past month6. Moreover, ACE scores of pregnant women have been linked to poor coping mechanisms such as illicit drug use during pregnancy7. These scores also impact prenatal, perinatal, and post-natal health8. For example, babies who were exposed to opioids in utero had significant associations with poorer health outcomes and delays in developmental stages9. Another study concluded that mothers suffering from substance use disorder engage in poor parenting practices such as "limited or absent parental monitoring and lower levels of parental involvement."10 Currently, many medical practices are using ACE scores as a general screening tool to help identify health risks and provide individualized care and family support11. Recent studies show that identifying positive childhood experiences is important when evaluating the impact of ACEs. Protective factors, such as resilience, can offset the negative health impacts of trauma12,13. Described as good outcomes in the face of a threat to wellbeing13, resilience can be quantified by using a questionnaire called the 7Cs tool14. The 7Cs tool, which examines an individual's competence, confidence, character, connection, contribution, coping and control, is a valid method to measure resilience. Currently, the 7Cs tool is internally validated for adolescents that have experienced trauma, and it has shown a correlation between better outcomes with a higher resilience score despite having higher ACE scores. Overall, there is limited information regarding ways to identify and determine the health impact of maternal resilience. More research is necessary to understand how ACEs and resilience affect postpartum outcomes in mothers with SUD and their child.

ELIGIBILITY:
Inclusion Criteria:

* Women between 12 weeks 0 days of pregnancy and 1 month postpartum AND 18 years and older

Exclusion Criteria:

* Women younger than 18 and/ or non-English speaking patients who cannot give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be English-speaking women between 12 weeks 0 days of pregnancy and
  1 month postpartum who are 18 years and older, and their child, newborn, or neonate (newborn) of uncertain viability who are being seen at Cooper University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Rate of Emergency Room Visits in the First Year of Life | At 12 months of age of the baby
  Emergency Room Visits over the first year will be evaluated at 12 months after the child's birth and will note the number of emergency room visits during the year.
Rate of adherence to AAP vaccination guideline in the First Year of Life | At 12 months of age of the baby
  Vaccination Adherence over the first year will be evaluated at 12 months after the child's birth and will note adherence to the AAP guideline for 2, 4, 6 month vaccines.

SECONDARY OUTCOMES:
Substance Use Program Continuation | Documentation will be evaluated at 12 months postpartum
  We will document if the mother continued with substance use treatment program as applicable
Custody of the child at discharge | At time of neonatal discharge
  We will document whether the biological mother was discharged from the hospital with custody of the child
Custody of the child at 12 month of life | Documentation will be evaluated at 12 months post-partum
  We will document whether the biological mother had custody of her child at 12 months post partum
Child development and growth over 2 years | Documentation will be evaluated at 12 and 24 months post-partum
  We will document the development and growth of the child of the mother filling out ACE information at at 12 and 24 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Abraham, Principal Investigator — Cooper Medical School of Rowan University; Hsiao-wei M Banks, Principal Investigator — Cooper Medical School of Rowan University
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellis MA, Hughes K, Leckenby N, Hardcastle KA, Perkins C, Lowey H. Measuring mortality and the burden of adult disease associated with adverse childhood experiences in England: a national survey. J Public Health (Oxf). 2015 Sep;37(3):445-54. doi: 10.1093/pubmed/fdu065. Epub 2014 Aug 30. PMID 25174044
- [Result] Exley D, Norman A, Hyland M. Adverse childhood experience and asthma onset: a systematic review. Eur Respir Rev. 2015 Jun;24(136):299-305. doi: 10.1183/16000617.00004114. PMID 26028641
- [Result] Su S, Wang X, Pollock JS, Treiber FA, Xu X, Snieder H, McCall WV, Stefanek M, Harshfield GA. Adverse childhood experiences and blood pressure trajectories from childhood to young adulthood: the Georgia stress and Heart study. Circulation. 2015 May 12;131(19):1674-81. doi: 10.1161/CIRCULATIONAHA.114.013104. Epub 2015 Apr 9. PMID 25858196
- [Result] Stein MD, Conti MT, Kenney S, Anderson BJ, Flori JN, Risi MM, Bailey GL. Adverse childhood experience effects on opioid use initiation, injection drug use, and overdose among persons with opioid use disorder. Drug Alcohol Depend. 2017 Oct 1;179:325-329. doi: 10.1016/j.drugalcdep.2017.07.007. Epub 2017 Aug 5. PMID 28841495
- See also: Related Info — https://www.samhsa.gov/data/sites/default/files/reports/rpt23250/5_Women_2020_01_14.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT05731557/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT05731557/ICF_001.pdf